CLINICAL TRIAL: NCT00792779
Title: Protective Effect of Propofol Against Hemolysis in Patients Submitted to Gastroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Medico Campinas (Other)
Responsible Party: Ricardo Francisco Simoni, Fundação Centro Médico de Campinas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE - 0023.0.263.000-08
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: Hemolysis
Keywords: Morbid obesity; General anaesthesia; Propofol; Sevoflurane
MeSH Terms: conditions — Hemolysis; Obesity, Morbid | interventions — Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Propofol — Patients in the Propofol Group (PG) will be induced with target-controlled infusion (TCI) of propofol (Diprifusor, AstraZeneca) and remifentanil (Asena PK, Cardinal Health) at the target dose of 6.0 µg.ml-1 and 8.0 ηg.ml-1, respectively. The patients in the Sevoflurane Group (SG) will be induced with remifentanil TCI at target dose of 8.0 ηg.ml-1 and etomidate 0.5 mg.kg-1 in bolus.

SUMMARY:
The purpose of this study is to determine if propofol could protect erythrocytes by directly scavenging free radicals from the blood current and increasing resistance of their cell membranes in patients submitted to gastroplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients between BMI 40-50 kg/m2

Exclusion Criteria:

* patients with BMI under 40 kg/m2 and over 50 kg/m2
* alcohol users
* illicit-drug users
* patients in regular use of anti-depressants, proton bomb inhibitors or calcium canal blockers
* patients transfused either recently, during the intra-operative period or within 10 hours post-operative
* patients previously known to be hypersensitive to any drug that is used during the study
* patients with any psychiatric disorder or dementia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-05 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Count erythrocytes | After 10 hours post-surgery

SECONDARY OUTCOMES:
Bilirubins(direct and indirect) | After 10 hours post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Simoni, MD, Principal Investigator — Fundação Centro Médico de Campinas
Locations (1):
- Fundação Centro Médico de Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Result] Tsuchiya M, Asada A, Kasahara E, Sato EF, Shindo M, Inoue M. Antioxidant protection of propofol and its recycling in erythrocyte membranes. Am J Respir Crit Care Med. 2002 Jan 1;165(1):54-60. doi: 10.1164/ajrccm.165.1.2010134. PMID 11779730